CLINICAL TRIAL: NCT01159275
Title: Pharmacokinetics of Pediatric Aluvia® (Lopinavir /Ritonavir 100/25 mg) and Generic Lopinavir/Ritonavir Tablet Formulation (200/50 mg) in Clinically and Virologically Stable HIV-1 Infected Thai Adults
Brief Title: Lopinavir (LPV) Dose Reduction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Ministry of Education, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HIV-NAT 085
Record Dates: First submitted 2010-06-04; First posted 2010-07-09 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV-1 Infections
Keywords: lopinavir/ritonavir; pharmacokinetics; HIV-1 infected adults; aim to investigate the lower dose of boosted lopinavir in Thais and to compare the levels of lopinavir/ritonavir from Abbot and GPO
MeSH Terms: interventions — lopinavir-ritonavir drug combination; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): First Generic LPV/r 200/50 mg BID, then cross over to Pediatric Aluvia 200/50 mg BID
  Interventions: Drug: Generic LPV/r and Aluvia (pharmacokinetics)
- 2 (Other): First Pediatric Aluvia® 200/50 mg BID, then cross over to Generic LPV/r 200/50 mg BID
  Interventions: Drug: Aluvia and Generic LPV/r (pharmacokinetics)

INTERVENTIONS:
Drug: Generic LPV/r and Aluvia (pharmacokinetics) — Generic LPV/r 200/50 mg BID 12 hr PK then cross over to Pediatric Aluvia 200/50 mg BID
  Arms: 1
Drug: Aluvia and Generic LPV/r (pharmacokinetics) — First Pediatric Aluvia® 200/50 mg BID, then cross over to Generic LPV/r 200/50 mg BID
  Arms: 2

SUMMARY:
The purpose of this study is to study the pharmacokinetics profiles of generic lopinavir/ritonavir and Pediatric Aluvia® at reduced dose by assessing safety, tolerability and efficacy.

DETAILED DESCRIPTION:
This is a prospective, 2 arms, randomized intensive PK study with cross over design. This design will provide us optimal information to answer our research question. First and most important, we can assess the PK when lopinavir/r is used in a dose reduced form. By randomizing the patients to either Abbott's pediatric Aluvia dose reduction or India generic LPV/r dose reduction will allow us to assess the differences in AE severity and frequency. Using the standard abbott product as a control our study will provide important information about the bioavailability of the generic product. Although it's not an original BE design we must be able to make preliminary comparisons.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Evidence of HIV infection (confirmed positive ELISA and/or documented history of measurable HIV RNA)
3. Age> 18 years
4. Have been on standard dose of any PI containing regimen for at least 4 weeks prior to study entry
5. Currently having no AIDS defining illness
6. Plasma HIV RNA < 50 copies/mL for at least 24 weeks
7. Willing to adhere to the protocol requirements

Exclusion Criteria:

1. Any history of taking CYP450 inhibitors or inducers, or any gastric acid-reducing drugs within 14 days of enrollment in the study
2. Current pregnancy or lactating
3. Active opportunistic infection
4. ALT/ AST more than 2x upper limit
5. creatinine more than 1.5 time the upper limit
6. Relevant history or current condition, illness that might interfere with drug absorption, distribution, metabolism or excretion
7. History of sensitivity/idiosyncrasy to the drug or chemically related compounds or pharmaceutical excipients which may be employed in the study.
8. Active drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
AUC, Cmin, Cmax of LPV/r between Aluvia and generic | week 2
  AUC, Cmin, Cmax of LPV/r between Aluvia and generic

CONTACTS AND LOCATIONS:
Overall Officials: Anchalee Avihingsanon, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration
Locations (1):
- HIV-NAT, Thai Red Cross AIDS Research Centre, Bangkok, Thailand

REFERENCES:
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org